CLINICAL TRIAL: NCT07173322
Title: The Impact of CAR-T Cell Therapy on Fertility; A Patient Survey
Status: Recruiting | Type: Observational
Sponsor: Blood Cancer United (Other)
Collaborators: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: LLSCART-25-001
Record Dates: First submitted 2025-08-29; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Cancer
Keywords: Cancer; CAR Tcell treatment
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
As there is limited knowledge regarding the impact of CAR-T Cell therapy on fertility, LLS has designed a Patient Survey to learn more about the impact on fertility in patients who have received/are receiving CAR-T Cell treatment. The insights gained from this survey will inform future treatment protocols and fertility preservation strategies.

ELIGIBILITY:
* any cancer patient
* at least 18 years of age
* with a history of receiving CAR-T Cell treatment.

less than 18 years old.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * any cancer patient
  * at least 18 years of age
  * with a history of receiving CAR-T Cell treatment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-02-09 (Actual); Primary Completion 2026-02-09 (Estimated); Study Completion 2026-02-09 (Estimated)

PRIMARY OUTCOMES:
The Impact of CAR-T Cell Therapy on Fertility | data will be collected for 1 year
  As there is limited knowledge regarding the impact of CAR-T Cell therapy on fertility, LLS, in collaboration with John Ligon MD and Citizen Health, has designed a Patient Survey to learn more about the impact on fertility in patients who have received/are receiving CAR-T Cell treatment. The insights gained from this survey will inform future treatment protocols and fertility preservation strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Nina Logan, MD, Principal Investigator — The Leukemia and Lymphoma Society; John J Ligon, MD, Study Chair — Univ of Florida, Gainesville
Locations (1):
- Internet, Rye, New York, United States

IPD SHARING:
Plan to Share IPD: No